CLINICAL TRIAL: NCT06622824
Title: Efficacy and Safety of Topical KX-826 Solution in Chinese Male Patients With Androgenetic Alopecia: A Multicenter, Randomized, Double-blind, Vehicle Controlled Adaptive Design Phase 2/3 Study
Brief Title: To Evaluate Efficacy and Safety of TopicalKX-826 Solution in Chinese Male Patients With Androgenetic Alopecia
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Suzhou Kintor Pharmaceutical Inc, (Industry)
Collaborators: Suzhou Koshine Biomedica, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KX0826-CN-1010
Record Dates: First submitted 2024-09-29; First posted 2024-10-02 (Actual); Last update posted 2024-10-21 (Actual); Status verified 2024-09

CONDITIONS: Androgenetic Alopecia (AGA)
Keywords: androgenetic alopecia; Hair loss
MeSH Terms: conditions — Alopecia | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A (Experimental): KX-826 0.5% BID
  Interventions: Drug: KX-826 0.5% BID
- Arm B (Experimental): KX-826 1.0% BID
  Interventions: Drug: KX-826 1.0% BID
- Arm C (Placebo Comparator): Matching Vehicle
  Interventions: Drug: Vehicle (Placebo) applied BID

INTERVENTIONS:
Drug: KX-826 0.5% BID — 0.5% of the investigational drug KX-826 to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm A
Drug: KX-826 1.0% BID — 1.0% of the investigational drug KX-826 to be applied topically to scalp twice daily for 24 weeks
  Arms: Arm B
Drug: Vehicle (Placebo) applied BID — Matching placebo applied topically to scalp twice daily for 24 weeks
  Arms: Arm C

SUMMARY:
This study is a multicenter, randomized, double-blind, vehicle controlled, adaptive design phase 2/3 study to evaluate the efficacy and safety of topical KX-826 solution in Chinese male patients with androgenetic alopecia (AGA). It consisted of two phases, phase 2 dose exploration trial and phase 3 confirmatory trial.

DETAILED DESCRIPTION:
In phase 2 study, around 90 adult male subjects with AGA (rating IIIv, IV and V on Hamilton-Norwood scale) were to be enrolled. All subjects would be evaluated with 1:1:1 randomized to receive KX-826 0.5% BID, KX-826 1.0% BID and vehicle in a double-blind fashion (30 subjects in each group), and would be treated for 24 weeks at the specified dose. During the study, the subjects would undergo periodic efficacy and safety-related examinations and evaluation. A Phase 2 statistical analysis will be performed when 90 patients complete the Week 24 visit or early withdrawal visit.

Blood samples will be collected at the following time points:

Day 1: 3 hours (pre-dose) W6 (Day 42): 3 hours (pre-dose) W12 (Day 84): 3 hours (pre-dose)

In phase 3 study, around 666 adult male subjects with AGA (rating IIIv, IV and V on Hamilton-Norwood scale) were to be enrolled. All subjects would be evaluated with 1:1:1 randomized to receive KX-826 0.5% BID, KX-826 1.0% BID and vehicle in a double-blind fashion (222 subjects in each group), and would be treated for 24 weeks at the specified dose. During the study, the subjects would undergo periodic efficacy and safety-related examinations and evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Agree to comply with study procedures and visit plan. Subject is capable of giving informed consent;
2. Male between the ages of 18 and 49 years, inclusive;
3. Clinically diagnosed as androgenetic alopecia;
4. Rating IIIv, IV and V on the Norwood Hamilton Scale; subject is willing to receive a ink dot tattoo;
5. Subject is willing to maintain the same hairstyle, hair length, and hair color at each visit;
6. Willing to use highly effective contraceptive measures during the study period and 3 months after the last dose.

Exclusion Criteria:

1. Had a history or active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania, or conditions/diseases other than AGA;
2. Had gray hair in the target alopecia area;
3. Had too short hair that, in the investogator's opinion, might affect hair growth assessment;
4. Had any skin pathology or condition that, in the investigator's opinion, could interfere with the evaluation of the investigational drug (e.g., fungal or bacterial infection, severe seborrheic dermatitis, solar keratosis, scalp psoriasis, contact dermatitis, severe folliculitis or scalp atrophy);
5. Had a significant increase in hair loss determined by investigator within 6 months prior to screening;
6. Had scalp hair transplants or hair extension history; need of wearing wig for a long time during the study;
7. Subjects who plan to use any adjuvant or concomitant therapy for the treatment of alopecia throughout the study;
8. Subjects with a previous or current diagnosis of hyperthyroidism or hypothyroidism;
9. Subjects with diseases that affect hair growth, such as connective tissue disease, inflammatory bowel disease, moderate to severe anemia, and significant short-term weight loss;
10. Had used finasteride or dutasteride prior to screening;
11. Had used platelet rich plasma (PRP) procedure within 12 months prior to screening;
12. Had used scalp surgical procedure within 12 months prior to screening; Had used laser, light, or energy treatments within 6 months of screening;
13. Had used anti-androgenic drugs (e.g., flutamide, cyproterone, drospirosterone, estrogen, progesterone, cimetidine, spironolactone, or oral ketoconazole, etc) within 6 months prior to screening;
14. Had used the following medications that may affect the evaluation of efficacy in the study within 6 months prior to screening:

    * Oral or topical minoxidil
    * Systemic interferon
    * Immunosuppressants such as cyclosporine
    * Diuretics
    * Beta-blockers (e.g., propranolol, atenolol, metoprolol, etc)
    * Anticoagulants (e.g., warfarin, heparin, heparin analogues, etc)
    * Anti-thyroid drugs (e.g., thiouracil, methiimidazole, etc)
    * Antipsychotic drugs (e.g., valproic acid, carbamazepine, phenytoin sodium, phenothiazines, fluoxetine, etc)
    * Anti-retroviral drugs (e.g., zidovudine, indonavir, ritonavir, lopinavir, etc)
    * Retinoids (e.g., actinoic acid, isotretinoic acid, etc), or use vitamin A supplements or A daily dietary intake of more than 10,000 IU of vitamin A
15. Used systemic steroids for more than 14 consecutive days within 3 months prior to screening;
16. Used oral hair growth supplements or herbs within 3 months prior to screening;
17. Use of hair growth shampoo such as ketoconazole or solution within 1 month prior to screening;
18. Subjects with acute infection of novel coronavirus and receiving (attenuated) live vaccine within 1 month prior to screening;
19. Abnormal and clinically significant findings in physical examination, vital signs, 12-lead ECG, hematology, urinalysis, blood chemistry, and thyroid function test at screening, which will affect the efficacy and safety evaluation and study results as judged by the investigator;
20. Positive blood screen for human immunodeficiency virus(HIV), hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody, or treponema pallidum antibody;
21. Have treated with KX-826 or GT20029 previously;
22. Subjects with sleep disorders, as assessed by the investigator, that affect hair growth, or the efficacy evaluation;
23. Subjects with depression, anxiety, or personality disorders, as assessed by the investigator, that affect hair growth, or the efficacy evaluation;
24. Has a known hypersensitivity or previous allergic reaction to any of the active or inactive ingredients in the investigational drug;
25. Medical/surgical history of any uncontrolled systemic disease that is serious or may affect the safety and efficacy evaluation of the investigational product, such as cardiovascular system, nervous system, hematological system, immune system, and psychiatric system disease;
26. Have undergone major surgery within 6 months prior to screening, or plan to undergo major surgery during the study;
27. Had a history of malignancy (except for cured carcinoma in situ) within 5 years prior to screening;
28. Subjects who have participated or are participating clinical studies of interventional drugs or medical devices within 3 months prior to screening;
29. Had a history of drug abuse within 12 months prior to screening;
30. Subjects who consumed large amounts of tea/coffee within 3 months prior to screening, as assessed by the investigator, that may affect hair growth, or the efficacy evaluation;
31. Subjects who, in the opinion of the investigator, have other conditions that may affect compliance or are not suitable for participation in this study;

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 756 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2027-10-20 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Target Area Non-vellus Hair count (TAHC) change from baseline at week 24 in comparison to vehicle. | 24 weeks
  Changes from baseline in non-vellus TAHC (Target Area Hair Counts) in comparison to vehicle (Non-vellus TAHC is the number of non-vellus hairs within 1 cm² scalp, which usually ranges from 0 to 300. Larger non-vellus TAHC implies thicker hair. In this study, larger change in non-vellus TAHC means better outcome.)

SECONDARY OUTCOMES:
Hair Growth Assessment (HGA) | 6 weeks, 12 weeks, 18 weeks and 24 weeks
  Changes from baseline HGA (Hair Growth Assessment) score by Principal Investigator and subjects (HGA scale ranged from -3 to 3 and represented decreases from baseline that were substantial, moderate, slight, no change, slight increases, moderate increases, and substantial increases, respectively. HGA improvement was defined as a hair growth assessment score of larger than 0.)
Target Area Non-vellus Hair diameter (TAHW) assessment | 6 weeks, 12 weeks, 18 weeks and 24 weeks
  Target Area Non-vellus Hair diameter (TAHW) change from baseline at week 6, 12, 18, and 24 in comparison to vehicle
Target Area total hair counts | 6 weeks, 12 weeks, 18 weeks and 24 weeks
  Target Area total hair counts change from baseline at week 6, 12, 18, and 24 in comparison to vehicle
TAHC assessment | 6 weeks, 12 weeks, 18 weeks
  Changes from baseline in non-vellus TAHC (Target Area Hair Counts) in comparison to vehicle (Non-vellus TAHC is the number of non-vellus hairs within 1 cm² scalp, which usually ranges from 0 to 300. Larger non-vellus TAHC implies thicker hair. In this study, larger change in non-vellus TAHC means better outcome.)

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No